CLINICAL TRIAL: NCT07097129
Title: Effect of Mask Ventilation on Surgical Field View in Robotic Colorectal Surgery: A Randomized Controlled Clinical Trial
Brief Title: Effect of Mask Ventilation on Surgical Field View in Robotic Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Kamil Darcin, MD, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024.286.IRB1.036
Record Dates: First submitted 2025-03-28; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Gastric Dilation; Bowel Distention; Surgical Procedure, Unspecified
Keywords: robotic colorectal surgery; gastric dilation; bowel distention; surgical view
MeSH Terms: conditions — Gastric Dilatation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The surgical team, who is blinded to the anaesthesia induction groups, will mark the Likert scale prepared for the presence of gastric distension, presence of intestinal distension, status of bowel movements and surgical vision regarding the intraoperative process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Mask Ventilation (Active Comparator): 2 mcg/kg fentanyl, 1 - 2 mg/kg propofol, 1 mg/kg rocuronium will be administered for anaesthesia induction. Orotracheal intubation will be performed at 60 seconds with video laryngoscopy without ventilation other than spontaneous breathing.
  Interventions: Procedure: Mask Ventilation
- Mask Ventilation (No Intervention): 2 mcg/kg fentanyl, 1 - 2 mg/kg propofol, 1 mg/kg rocuronium will be administered for anaesthesia induction. Mask ventilation will be performed with mechanical ventilator set to pressure controlled ventilation, 15 cmH20 peak pressure, 10 respiratory rates per minute. Orotracheal intubation will be performed at the 60th second with video laryngoscopy.

INTERVENTIONS:
Procedure: Mask Ventilation — Mask ventilation with mechanical ventilator set to pressure controlled ventilation, 15 cmH20 peak pressure, 10 respiratory rates per minute
  Arms: No Mask Ventilation

SUMMARY:
The goal of this clinical trial is to demonstrate the effects of pressure-controlled mask ventilation and non-mask ventilation during anaesthesia induction on gastric insufflation, gastric dilatation, increased bowel movements and bowel distension and to demonstrate its effect on surgical vision in robotic colorectal surgeries. The main questions it aims to answer are:

How will non-mask ventilation during anaesthesia induction effect surgical vision in robotic colorectal surgeries compared to mask ventilation? How will non-mask ventilation during anaesthesia induction effect gastric dilatation and bowel movements in robotic colorectal surgeries compared to mask ventilation?

If there is a comparison group: Researchers will compare mask ventilation and non-mask ventilation during anaesthesia induction to see if the surgical vision, gastric dilatation and bowel movements are effected.

Participants will be divided in two groups:

No mask ventilation group: Outside of spontaneous breathing during preoxygenation, orotracheal intubation will be performed at the 60th second after anesthesia induction without ventilation, using video laryngoscopy. Mask ventilation group: After anesthesia induction, mask ventilation will be performed with a respiratory rate of 10 and 15 cmH2O pressure, followed by orotracheal intubation using video laryngoscopy at the 60th second.

Researchers will compare the results between the groups to see the surgical vision, gastric dilatation and bowel movements.

The hypothesis of this study is that non-mask ventilation will provide better surgical vision, less gastric dilatation and less bowel movements in robotic colorectal surgeries.

DETAILED DESCRIPTION:
Following anaesthesia induction, mask ventilation is a technique applied until successful tracheal intubation is achieved. It is known that with mask ventilation, air can also enter the stomach as well as the trachea. If mask ventilation is not performed with the correct technique during robotic surgery, excessive dilation of the stomach will impair the surgical team's vision, causing the operation to be more difficult and longer. In this study, we aimed to demonstrate the effects of mask ventilation and non-mask ventilation on gastric dilatation, increased bowel movements, bowel distension and surgical vision in robotic colorectal surgeries.

In our anaesthesia practice, patients will be premedicated with 0.03 mg/kg midazolam in the preoperative area and then taken to the operating room. After standard monitorization in the operating room, preoxygenation will be applied with end tidal oxygen (EtO2) monitoring. Patients whose EtO2 value reached 90% will be divided into two groups and the following protocol will be applied; No mask ventilation group: 2 mcg/kg fentanyl, 1 - 2 mg/kg propofol, 1 mg/kg rocuronium will be administered for anaesthesia induction. Orotracheal intubation will be performed at 60 seconds with video laryngoscopy without ventilation other than spontaneous breathing.

Mask ventilation group: 2 mcg/kg fentanyl, 1 - 2 mg/kg propofol, 1 mg/kg rocuronium will be administered for anesthesia induction. Mask ventilation will be performed with mechanical ventilator set to pressure controlled ventilation, 15 cmH20 peak pressure, 10 respiratory rates per minute. Orotracheal intubation will be performed at the 60th second with video laryngoscopy.

The surgical team, who is blinded to the anesthesia induction groups, will mark the Likert scale prepared for the presence of gastric distension, presence of intestinal distension, status of bowel movements and surgical vision regarding the intraoperative process. Surgical time will also be recorded at the end of the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 80 who are scheduled to undergo robotic colorectal surgery will be included in the study.

Exclusion Criteria:

* Patients with preoperative prediction of possible difficult intubation
* Presence of restrictive/obstructive lung disease requiring CPAP application for treatment in preoperative anaesthesia evaluation
* Patients with cardiovascular diseases (EF < 20%, advanced aortic stenosis, decompensated heart failure) that require change of at least one of the drugs to be used for anaesthesia induction
* Presence of allergy to any of the drugs to be used in anaesthesia induction and maintenance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Surgical Vision | 5 minutes after the end of the surgical procedure
  Likert scale Surgical field visibility is very poor: 1 point Surgical field visibility is poor: 2 points Surgical field visibility is moderate: 3 points Surgical field visibility is good: 4 points Surgical field visibility is very good: 5 points
  Higher scores on this scale mean a better outcome.
Gastric Dilatation | 5 minutes after the end of the surgical procedure
  Likert Scale Gastric dilatation was severe enough to complicate the surgical technique: 1 point Gastric dilatation was present but did not complicate the surgery: 2 points Stomach was not dilated: 3 points
  Higher scores on this scale mean a better outcome.
Bowel distension | 5 minutes after the end of the surgical procedure
  Likert Scale Bowel distension is quite significant: 1 point Bowel distension is significant: 2 points Bowel distension is moderate: 3 points Bowel distension is mild: 4 points No bowel distension: 5 points
  Higher scores on this scale mean a better outcome.
Bowel movement | 5 minutes after the end of the surgical procedure
  Likert Scale Bowel movements are quite frequent: 1 point Bowel movements are frequent: 2 points Bowel movements are moderate: 3 points Bowel movements are mild: 4 points No bowel movements: 5 points
  Higher scores on this scale mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Koç University Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting from 6 months after publication for 5 years
Access Criteria: No access criteria

REFERENCES:
- [Background] Jung YK, Kim CL, Jeong MA, Sung JM, Lee KG, Kim NY, Kang L, Lim H. Gastric insufflation and surgical view according to mask ventilation method for laparoscopic cholecystectomy: a randomized controlled study. BMC Anesthesiol. 2023 Sep 20;23(1):321. doi: 10.1186/s12871-023-02269-9. PMID 37730575
- [Background] Bouvet L, Albert ML, Augris C, Boselli E, Ecochard R, Rabilloud M, Chassard D, Allaouchiche B. Real-time detection of gastric insufflation related to facemask pressure-controlled ventilation using ultrasonography of the antrum and epigastric auscultation in nonparalyzed patients: a prospective, randomized, double-blind study. Anesthesiology. 2014 Feb;120(2):326-34. doi: 10.1097/ALN.0000000000000094. PMID 24317204